CLINICAL TRIAL: NCT03561961
Title: Randomised Controlled Trial of Prostate Radiotherapy In High Risk and Node Positive Disease Comparing Moderate and Extreme Hypo-fractionation (PRIME Trial)
Brief Title: Prostate Radiotherapy Comparing Moderate and Extreme Hypo-fractionation (PRIME Trial)
Acronym: PRIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Collaborators: Tata Medical Center (Other)
Responsible Party: Principal Investigator, Dr Vedang Murthy, Professor, Radiation Oncology, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRIME
Record Dates: First submitted 2018-05-23; First posted 2018-06-19 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Hypo-fractionation (Active Comparator): In arm 1 of the study, patients who are randomized to receive moderately hypo-fractionated RT will receive a total dose of 66-68 Gy in 25# to the primary over 5 weeks, with treatment being delivered daily. All patients will receive a dose of 50 Gy in 25# to the pelvis. Boost to gross nodal disease will be considered based on the response to hormonal therapy to a dose of 60-66 Gy/25# as a simultaneous integrated boost(SIB).
  Interventions: Radiation: Moderate Hypo-fractionation
- Extreme Hypo-fractionation (Experimental): In Arm 2 of the study, patients who are scheduled to receive SBRT will receive a course of 5 fractions of radiation; each fraction size will be 7.00-7.25 Gy. The total dose will be 35-36.5 Gy. All patients will receive a dose of 25 Gy in 5 # to the pelvis. Boost to gross nodal disease will be considered based on the response to hormonal therapy to a dose of 30-35 Gy/5# as a simultaneous integrated boost(SIB).The 5 treatments will be scheduled to be delivered alternate day over approximately 7-10 days. An option of equivalent biological dose using 35-36.5 Gy in 5 weekly fractions may be allowed for multicentric accrual in the future.
  Interventions: Radiation: Extreme Hypo-fractionation

INTERVENTIONS:
Radiation: Moderate Hypo-fractionation — 66-68Gy in 25#
  Arms: Moderate Hypo-fractionation
Radiation: Extreme Hypo-fractionation — 35-36.25 Gy in 5#
  Other Names: SBRT
  Arms: Extreme Hypo-fractionation

SUMMARY:
Aim: The aim of the study is to compare the efficacy with SBRT and moderate hypo-fractionation in high risk and node positive prostate cancer

PRIMARY STUDY OBJECTIVES: To assess whether extreme hypo-fractionation with SBRT in high risk prostate cancer is non inferior to moderately hypo-fractionated standard radiotherapy

STUDY DESIGN: Two arm, Prospective Randomized Trial with a non-inferiority design

TREATMENT REGIMEN: Arm 1-[standard arm] Moderate hypo-fractionated RT, total dose of 66-68 Gray(Gy) in 25# to the primary over 5 weeks, with treatment being delivered daily. All patients irrespective of nodal status will receive a dose of 50 Gy in 25# to the pelvic nodes.Boost to gross nodal disease will be considered based on the response to hormonal therapy to a dose of 60-66 Gy/25# as a simultaneous integrated boost (SIB). An option of equivalent biological dose using 60-62.5 Gy in 20# may be allowed for multi-centric accrual in the future.

Arm 2 -[Experimental Arm] Extreme hypo-fractionation with SBRT,course of 5 fractions of radiation; each of size 7-7.25 Gy. The total dose will be 35-36.5 Gy. All patients irrespective of nodal status will receive a dose of 25 Gy in 5 # to the pelvic nodes. The 5 treatments will be scheduled to be delivered alternate day over approximately 7-10 days. An option of equivalent biological dose using 35-36.5 Gy in 5 weekly fractions may be allowed for multicentric accrual in the future.

RECRUITMENT TARGET: 464 total (232 patients experimental arm and 232 patients standard arm) recruitment over 6 years, with a non-fixed follow up period and a uniform accrual rate.

PRIMARY ENDPOINT To assess the 5 year Biochemical Failure free Survival (BFFS) between the two arms.

Follow-up At 3-6 weeks from end of radiotherapy, followed by 3-6 monthly for the first two years and 6 monthly thereafter.

DETAILED DESCRIPTION:
The standard duration of treatment with radiotherapy is 8 weeks in conventional fractionation; 5-6 weeks with moderate hypo-fractionation, while it is only 1- 2 weeks with extreme hypo-fractionation (SBRT).The health costs and out of pocket expenditure involved in the conventional hypo-fractionated radiotherapy treatment largely depends on the overall treatment duration. This involves expenditure not only for the patient but also the caretaker. Moreover most of these patients presenting to a tertiary care centre from different parts of the country, have logistic issues of accommodation, food, travel along with the treatment costs. Also for patients staying away from family, 5 weeks treatment without considerable family support has a psychological impact, especially on elderly group of patients commonly seen with prostate cancer.This further leads to a major cause of distress among these patients, especially in a resource limited setting as ours.

Extreme hypo-fractionation with a total duration of 2 weeks, would offer an opportunity to optimize the therapeutic ratio taking advantage of the potential therapeutic gain due to low alpha/beta for prostate to higher dose/fraction(compared to surrounding organs at risk). Moreover, shortened overall treatment time,would lead to less distressing and early recommencement of their daily activities for the patients,with an obvious impact in improving the quality of life and health costs.

Given the potential positive economic impact with shorter duration treatment with similar clinical outcomes and probable similar toxicity profile, SBRT (extreme hypo-fractionation) in prostate cancer is an attractive treatment option, especially in a limited-resource setting and can have a large and positive impact on the patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Age: above 18 years.
2. Participants must be histologically proven, adenocarcinoma prostate
3. Localised to the prostate or pelvic lymph nodes
4. High risk prostate cancer as defined by National Comprehensive Cancer Network (NCCN):Gleason score of 8-10, clinical stage T3a or higher, or PSA > 20 ng/mL.
5. Ability to receive long term hormone therapy/ orchidectomy
6. Karnofsky Performance Score (KPS) >70 (see appendix
7. No prior history of therapeutic irradiation to pelvis
8. Patient willing and reliable for follow-up and QOL.
9. Signed study specific consent form

Exclusion Criteria:

1. Evidence of distant metastasis at any time since presentation
2. Life expectancy <2 year
3. Previous RT to prostate or prostatectomy.
4. A previous trans-urethral resection of the prostate (TURP)
5. Severe urinary symptoms or with severe International Prostate Symptom Score (IPSS) score despite being on hormonal therapy for 6 months which in the opinion of the physician precludes RT
6. Patients with known obstructive symptoms with stricture.
7. Any contraindication to radiotherapy like inflammatory bowel disease.
8. Uncontrolled comorbidities including, but not limited to diabetes or hypertension
9. Unable to follow up or poor logistic or social support

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2035-03 (Estimated)

PRIMARY OUTCOMES:
Biochemical Failure free Survival (BFFS) | 5 years
  Freedom from biochemical failure will be defined as duration from date of nadir Prostate Specific Antigen (PSA) to PSA>2ng/ml over the nadir PSA

SECONDARY OUTCOMES:
Acute toxicity with both treatments. | 2 years
  Radiation Therapy Oncology Group (RTOG) and CTCAE v 4
Late toxicity with both treatments. | 2 years
  Radiation Therapy Oncology Group (RTOG) and CTCAE v 4
Prostate cancer specific survival | 5 years
  calculated from the date of randomization to the date of the death due to prostate cancer
Overall Survival | 5 years
  defined as the time from randomization to the time of death from any cause
out of pocket expenditure | Baseline, 2 and 5 years
  structured case record form
patient reported quality of life | baseline and every 6 monthly for five years
  EORTC Quality of Life Questionnaire Core 30 (QLQc30) and Prostate 25 (PR25)

CONTACTS AND LOCATIONS:
Overall Officials: Vedang Murthy, Principal Investigator — Tata Memorial Centre
Locations (1):
- Dr Vedang Murthy, Navi Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murthy V, Mallick I, Gavarraju A, Sinha S, Krishnatry R, Telkhade T, Moses A, Kannan S, Prakash G, Pal M, Menon S, Popat P, Rangarajan V, Agarwal A, Kulkarni S, Bakshi G. Study protocol of a randomised controlled trial of prostate radiotherapy in high-risk and node-positive disease comparing moderate and extreme hypofractionation (PRIME TRIAL). BMJ Open. 2020 Feb 28;10(2):e034623. doi: 10.1136/bmjopen-2019-034623. PMID 32114475
- See also: Acute toxicity — https://doi.org/10.1016/S0167-8140(23)08750-9

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT03561961/Prot_SAP_000.pdf